CLINICAL TRIAL: NCT06694727
Title: A Danish Pragmatic Randomized Trial of Nutritional Supplements in Heart Failure (DANUTRIO-HF: Q10, DANUTRIO-HF: Selenium)
Brief Title: A Danish Pragmatic Randomized Trial of Nutritional Supplements in Heart Failure
Acronym: DANUTRIO-HF
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tor Biering-Sørensen (Other)
Collaborators: Pharma Nord (Industry)
Responsible Party: Sponsor-Investigator, Tor Biering-Sørensen, Professor, MD, MSc, MPH, PhD, Herlev and Gentofte Hospital
Organization: Herlev and Gentofte Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DANUTRIO-HF
Record Dates: First submitted 2024-10-28; First posted 2024-11-19 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure
Keywords: Heart failure; Coenzyme Q10; Selenium; Randomized Controlled Trial; Registry; Echocardiography; Pragmatic; Factorial; 2x2; Cardiovascular; Nutritional supplements
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 fashion to receive either the experimental intervention or placebo for each of the two nutritional supplements.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Coenzyme Q10 intervention, active (Experimental): 100 mg capsules given twice daily, per oral use
  Interventions: Dietary Supplement: Coenzyme Q10 100 Milligrams Oral Capsule
- Coenzyme Q10 intervention, placebo (Placebo Comparator): Placebo matching coenzyme Q10
  Interventions: Dietary Supplement: Coenzyme Q10 100 Milligrams Oral Capsule
- Selenium intervention, active (Experimental): 100 μg tables given twice daily, per oral use
  Interventions: Dietary Supplement: Selenium 100 Micrograms Oral Tablets
- Selenium intervention, placebo (Placebo Comparator): 100 μg tables given twice daily, per oral use
  Interventions: Dietary Supplement: Selenium 100 Micrograms Oral Tablets

INTERVENTIONS:
Dietary Supplement: Coenzyme Q10 100 Milligrams Oral Capsule — 100 mg capsules given twice daily, per oral use.
  Arms: Coenzyme Q10 intervention, active; Coenzyme Q10 intervention, placebo
Dietary Supplement: Selenium 100 Micrograms Oral Tablets — 100 μg tablets given twice daily, per oral use.
  Arms: Selenium intervention, active; Selenium intervention, placebo

SUMMARY:
Heart failure is a common and serious condition. Despite rapid advancements in heart failure treatment, the prognosis remains severe. Smaller studies have shown that two simple, safe, and relatively inexpensive nutritional supplements-coenzyme Q10 and selenium-may reduce the risk of complications associated with heart failure. The DANUTRIO-HF trial will investigate whether these supplements can make a difference for individuals with heart failure. The study will assign approximately 4,044 patients from across Denmark to either coenzyme Q10 (100 mg twice daily) or a corresponding placebo, as well as selenium (100 μg twice daily) or its corresponding placebo, and follow how many of them end up being hospitalized for heart failure or dying from heart problems over an estimated two to three-year period.

DETAILED DESCRIPTION:
This investigator-initiated, pragmatic, registry-based, double-blinded, placebo-controlled, 2x2 factorial, individually randomized trial aims to evaluate the efficacy of daily intake of the nutritional supplements coenzyme Q10 versus placebo, and selenium versus placebo, in preventing heart failure hospitalizations and cardiovascular death in heart failure patients. The trial plans to randomize approximately 4,044 participants in an event-driven design. Participants will be identified through the Danish Administrative Health Registries, which will also serve as the primary source for data collection. Contact with potential participants will be made via the mandatory Danish electronic letter system. No scheduled in-person visits are required in the main study, and all study interventions will be mailed to participants.

A substudy involving up to 600 participants will assess the effects of coenzyme Q10 and selenium on functional capacity, treatment compliance, biochemical biomarkers, and cardiac function and structure. This group will attend two in-person visits for additional evaluations, including echocardiography, blood sampling, and a 6-minute walk test at baseline and at the 1-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged ≥ 18 years.
* Registered with a heart failure diagnosis (ICD-10: I50) as a primary discharge diagnosis in The Danish National Patient Registry and at least one claimed prescription of a renin-angiotensin-system inhibitor and a β-blocker within 120 days after HF diagnosis.
* Informed consent form has been signed and dated.

Exclusion Criteria:

* Use of vitamin K-antagonist
* Registered with a cancer diagnosis (C00-C97 not C44) within the last 5 years excluding cutaneous squamous cell or basal cell carcinoma in The Danish National Patient Registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4044 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Time to the first occurrence of hospitalization for heart failure or cardiovascular death | From date of randomization until end of study (Up to approximately 33 months)

SECONDARY OUTCOMES:
Time to first occurrence of hospitalization for heart failure | From date of randomization until end of study (Up to approximately 33 months)
Time to cardiovascular death | From date of randomization until end of study (Up to approximately 33 months)

OTHER OUTCOMES:
Total number of hospitalizations for heart failure | From date of randomization until end of study (Up to approximately 33 months)
Total number of hospitalizations for heart failure and cardiovascular death | From date of randomization until end of study (Up to approximately 33 months)
Time to the first occurrence of hospitalization for heart failure or all-cause death | From date of randomization until end of study (Up to approximately 33 months)
Total number of hospitalizations for heart failure and all-cause death | From date of randomization until end of study (Up to approximately 33 months)
Time to all-cause mortality | From date of randomization until end of study (Up to approximately 33 months)
Time to first occurrence of major adverse cardiovascular events | From date of randomization until end of study (Up to approximately 33 months)
Total number of major adverse cardiovascular events | From date of randomization until end of study (Up to approximately 33 months)
Time to first occurrence of hospitalization for any cardiovascular disease | From date of randomization until end of study (Up to approximately 33 months)
Total number of hospitalizations for any cardiovascular disease | From date of randomization until end of study (Up to approximately 33 months)
Time to first occurrence of hospitalization for any cardiorespiratory disease | From date of randomization until end of study (Up to approximately 33 months)
Total number of hospitalizations for any cardiorespiratory disease | From date of randomization until end of study (Up to approximately 33 months)
Time to first hospitalization for atrial fibrillation | From date of randomization until end of study (Up to approximately 33 months)
Total number of hospitalizations for atrial fibrillation | From date of randomization until end of study (Up to approximately 33 months)
Time to first occurrence of hospitalization for cardiac arrest | From date of randomization until end of study (Up to approximately 33 months)
Time to first hospitalization for any cause | From date of randomization until end of study (Up to approximately 33 months)
Total number of hospitalizations for any cause | From date of randomization until end of study (Up to approximately 33 months)
Change in Kansas City Cardiomyopathy Questionnaire Score | Aproximately within 1 year after randomization
Change in left ventricular ejection fraction assessed with echocardiography | Aproximately within 1 year after randomization
  In up to 600 participants in a planned substudy with two physical visits. One shortly after randomization and another 1 year after
Change in left ventricular global longitudinal strain assessed with echocardiography | Aproximately within 1 year after randomization
  In up to 600 participants in a planned substudy with two physical visits. One shortly after randomization and another 1 year after
Change in E/e'-ratio assessed with echocardiography | Aproximately within 1 year after randomization
  In up to 600 participants in a planned substudy with two physical visits. One shortly after randomization and another 1 year after
Change in left ventricular mass assessed with echocardiography | Aproximately within 1 year after randomization
  In up to 600 participants in a planned substudy with two physical visits. One shortly after randomization and another 1 year after
Change in interventricular septal wall thickness assessed with echocardiography | Aproximately within 1 year after randomization
  In up to 600 participants in a planned substudy with two physical visits. One shortly after randomization and another 1 year after
Change in left ventricular posterior thickness assessed with echocardiography | Aproximately within 1 year after randomization
  In up to 600 participants in a planned substudy with two physical visits. One shortly after randomization and another 1 year after
Change in left atrial volume assessed with echocardiography | Aproximately within 1 year after randomization
  In up to 600 participants in a planned substudy with two physical visits. One shortly after randomization and another 1 year after
Change in left atrial resevoir strain assessed with echocardiography | Aproximately within 1 year after randomization
  In up to 600 participants in a planned substudy with two physical visits. One shortly after randomization and another 1 year after
Change in left atrial contraction strain assessed with echocardiography | Aproximately within 1 year after randomization
  In up to 600 participants in a planned substudy with two physical visits. One shortly after randomization and another 1 year after
Change in left atrial conduit strain assessed with echocardiography | Aproximately within 1 year after randomization
  In up to 600 participants in a planned substudy with two physical visits. One shortly after randomization and another 1 year after
Change in tricuspid annular plane systolic excursion assessed with echocardiography | Aproximately within 1 year after randomization
  In up to 600 participants in a planned substudy with two physical visits. One shortly after randomization and another 1 year after
Change in right ventricular free wall longitudinal strain assessed with echocardiography | Aproximately within 1 year after randomization
  In up to 600 participants in a planned substudy with two physical visits. One shortly after randomization and another 1 year after
Change in pro-BNP | Aproximately within 1 year after randomization
  In up to 600 participants in a planned substudy with two physical visits. One shortly after randomization and another 1 year after
Change in high sensitivity troponin-I | Aproximately within 1 year after randomization
  In up to 600 participants in a planned substudy with two physical visits. One shortly after randomization and another 1 year after
Change in hs-CRP | Aproximately within 1 year after randomization
  In up to 600 participants in a planned substudy with two physical visits. One shortly after randomization and another 1 year after
Concentration of coenzyme Q10 at followup | Aproximately within 1 year after randomization
  In up to 600 participants in a planned substudy with two physical visits. One shortly after randomization and another 1 year after
Concentration of selenoprotein P and selenium at followup | Aproximately within 1 year after randomization
  In up to 600 participants in a planned substudy with two physical visits. One shortly after randomization and another 1 year after
Change in 6 minute walking distance | Aproximately within 1 year after randomization
  In up to 600 participants in a planned substudy with two physical visits. One shortly after randomization and another 1 year after

CONTACTS AND LOCATIONS:
Overall Officials: Tor Biering-Sørensen, MD, MPH, MSc, PhD, Principal Investigator — Center for Translational Cardiology and Pragmatic Randomized Trials, Department of Cardiology, Copenhagen University Hospital - Herlev and Gentofte
Locations (1):
- Center for Translational Cardiology and Pragmatic Randomized Trials, Department of Cardiology, Copenhagen University Hospital - Herlev and Gentofte, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Most data will be collected from Danish administrative health registries, which are subject to Danish legislation and can only be made available to a third party under certain conditions. Please contact the sponsor-investigator in case of any inquiries.
Supporting Information: Study Protocol, SAP